CLINICAL TRIAL: NCT04696328
Title: Clinical Trial of Human (Allogeneic) iPS Cell-derived Cardiomyocytes Sheet for Ischemic
Brief Title: Clinical Trial of Human (Allogeneic) iPS Cell-derived Cardiomyocytes Sheet for Ischemic Cardiomyopathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Cuorips Inc. (Unknown)
Responsible Party: Principal Investigator, Koichi Toda, Associate Professor, Osaka University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVSC0005
Record Dates: First submitted 2020-12-11; First posted 2021-01-06 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Myocardial Ischemia
Keywords: ischemic cardiomyopathy, D017202
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group of subjects undergoing cell transplantation (Experimental): Human (allogeneic) iPS cell derived-cardiomyocyte sheet transplantation (only once)
  Interventions: Biological: Human (allogeneic) iPS cell derived-cardiomyocyte sheet

INTERVENTIONS:
Biological: Human (allogeneic) iPS cell derived-cardiomyocyte sheet — Transplantation

SUMMARY:
Targeting patients with severe ischemic cardiomyopathy, the purpose of this study is as follows: to confirm short-term efficacy by observing changes and transitions in cardiac function and clinical symptoms compared with each patient's baseline (before and after comparison) by human iPS cell-derived cardiomyocyte sheet transplantation, and to evaluate the safety and tolerability including the combined use of immunosuppressants.

DETAILED DESCRIPTION:
The objective of this study is to confirm the efficacy and safety of a human (allogeneic) iPS cell-derived cardiomyocyte sheet in combination with an immunosuppressant for ischemic cardiomyopathy patients. The primary evaluation items will be improvement of left ventricular systolic function (LVEF) for efficacy, and safety will be assessed by blood tests, general laboratory tests, and other safety-related evaluations. Secondary evaluation items are NYHA functional evaluation, left ventricular remodeling evaluation by echocardiography, hemodynamic evaluation, physical activity function evaluation such as 6MWD and SAS, QOL, and exercise tolerance evaluation by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic ischemic heart disease
2. Patients with Grade III-IV NYHA Functional Classification heart failure
3. Patients who are in the state of heart failure despite maximal oral medications including digitalis, diuretics, ACE inhibitors, ARBs, beta-blockers, anti-aldosterone drugs, and oral cardiotonics
4. Patients who are 20 years of age or older at the point of consent
5. Patients at risk of worsening heart failure despite being under standard surgical treatment (coronary artery bypass surgery, mitral valve angioplasty, left ventricular angioplasty, cardiac resynchronization therapy, and percutaneous coronary intervention) for more than 3 months
6. Patients with LVEF (Echocardiography) at rest of 35% or less
7. Patients whose informed consent for clinical trial participation can be obtained from the subject himself/herself in writing
8. Patients who can continue to visit to the clinical trial site for 52 weeks after obtaining consent, continue to live in Japan, and can be expected to have data collected by NRMD/PMS

Exclusion Criteria:

1. Patients with autoimmune diseases
2. Patients with allergies or hypersensitivity to the immunosuppressant used
3. Patients with active infections
4. Patients who remain in shock due to worsening heart failure
5. Patients with irreversible organ failure other than heart
6. Patients with malignant tumors
7. Patients who are or may be pregnant
8. Patients with history of alcoholism or drug addiction within six months from the day of consent
9. Patients with allergies or hypersensitivity to animals such as cattle from which the raw materials are derived
10. Patients with severe pulmonary hypertension
11. Patients within 6 months of completion of other clinical trials at the time of enrollment
12. In addition, patients with other cardiovascular abnormalities who are determined to be unfit for this study as per the judgment of the patient enrollment study committee of physicians

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
The number of patients with improved LVEF | 26 weeks
  The number of patients with improved LVEF by echocardiography 26 weeks postoperatively compared with preoperatively.
Incidence of adverse events and defects [Safety and Tolerability] | From postoperative to the end of the observation period (52 weeks)
  Regarding adverse events and side effects (of the adverse events, those whose causal relationship with the clinical trial product is determined to be other than "not related" will be treated as side effects.) the number of occurrences and the number of occurrence examples by event and severity will be obtained.
Incidence of serious adverse events [Safety and Tolerability] | From postoperative to the end of the observation period (52 weeks)
  Regarding serious adverse events, the number of occurrences and the number of occurrence examples by event and severity will be obtained.
Incidence of abnormal vital signs [Safety and Tolerability] | Before surgery, 7 days, 14 days, 4 weeks, 13 weeks, 26 weeks, 52 weeks
  Regarding changes in vital signs(Body temperature, blood pressure (systolic, diastolic), and pulse rate), summary statistics and changes at each measurement time point will be obtained.
Incidence of abnormal general blood tests [Safety and Tolerability] | Before surgery, 1 days, 7 days, 14 days, 4 weeks, 13 weeks, 26 weeks, 52 weeks
  Regarding changes in general blood tests(WBC, RBC, Hb, Ht, PLT), summary statistics and changes at each measurement time point will be obtained.
Incidence of abnormal blood biochemical tests [Safety and Tolerability] | Before surgery, 1 days, 7 days, 14 days, 4 weeks, 13 weeks, 26 weeks, 52 weeks
  Regarding changes in blood biochemistry tests(AST(GOT), ALT(GPT), LDH, ALP, BUN, Cre, UA, TG, T-Cho, LDL-Cho, Alb, CK, CK-MB, electrolytes (Na, K, Cl, Ca, iP, Mg), CRP, blood sugar), summary statistics and changes at each measurement time point will be obtained.
Incidence of abnormal tumor marker tests [Safety and Tolerability] | Screening, 13 weeks, 26 weeks, 52 weeks
  Regarding changes in tumor marker tests(AFP, CA19-9, CEA, hCG), summary statistics and changes at each measurement time point will be obtained.
Incidence of cardiac function clinical events such as death and hospitalization [Safety and Tolerability] | From postoperative to the end of the observation period (52 weeks)
  With respect to the incidence of cardiac function clinical events such as death and hospitalization, the number of cases in which the causes of death are related to heart disease and those unrelated to heart disease will be determined for cases of death.

SECONDARY OUTCOMES:
Number of Responder patients 26 and 52 weeks after transplantation of this product | 26 and 52 weeks
  To comprehensively evaluate the efficacy of this product transplantation
Contraction function of the entire left ventricle | 26 weeks
  To comprehensively evaluate the efficacy of this product transplantation
Left ventricular remodeling (LVESVI) | 26 weeks
  Changes in left ventricular end systolic volume index (LVESVI) (echocardiography, CT (if available))
Left ventricular remodeling (LVEDVI) | 26 weeks
  Changes in left ventricular end-diastolic volume index (LVEDVI) (echocardiography, CT (if available))
New York Heart Association functional classification | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. Class I to Class IV, the more severe, the higher the number.
Specific Activity Scale (SAS) | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. This is a quantitative evaluation of the subjective symptoms of heart failure from the viewpoint of exercise tolerance. List various daily activities for which exercise intensity [oxygen uptake or metabolic equivalents (METs)] is almost known in advance, ask whether they are possible, and exercise with the lowest activity level that was not possible is evaluated value. The higher the number, the better the condition.
The Minnesota Living with Heart Failure Questionnaire | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. The lower the number, the better the condition.
36-Item Short Form Survey (SF-36) | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. The higher the number, the better the condition.
6-minute walking distance | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. The higher the number, the better the condition.
Brain natriuretic peptide (BNP) | Before surgery, 1 days, 7 days, 14 days, 4 weeks, 13 weeks, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions.
N-terminal pro-brain natriuretic peptide (NT-proBNP) | Before surgery, 1 days, 7 days, 14 days, 4 weeks, 13 weeks, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions.
Exercise tolerance (VO2max) | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. Measure the maximum oxygen uptake (VO2max) using the bicycle ergometer.
Exercise tolerance (AT) | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. Measure the anaerobic metabolism threshold (AT) using the bicycle ergometer.
Exercise tolerance (VE/VCO2) | Before surgery, 26 weeks, 52 weeks
  Evaluation of the following changes and transitions before and 26 and 52 weeks after surgery. Measure the expiratory minute volume (VE)/the CO2 uptake (VCO2) using the bicycle ergometer.
Cumulative number of rejections that occurred during the observation period | 26 weeks
  Cumulative number of rejections from transplant up to 26 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiki Sawa, Ph.D, Study Director — Osaka University
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
Not planned at this time.